CLINICAL TRIAL: NCT04045743
Title: Clinical Efficacy of Inhibition of Organ Dysfunction Through Bermekimab in Systemic Sclerosis: A Proof- Of-Concept Double-Blind Randomized Clinical Trial (the Light Trial)
Brief Title: The Benefit of Bermekimab in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIGHT
Record Dates: First submitted 2019-07-27; First posted 2019-08-06 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2021-01

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — bermekimab

STUDY DESIGN:
Intervention Model Description: Patients assigned to either subcutaneous Bermekimab or placebo for 12 weeks ( 1:1 randomization, blind period ), then all patients are assigned to subcutaneous Bermekimab for 12 weeks ( open label period )
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bermekimab (MABp1) (Experimental)
  Interventions: Drug: MABp1 (Bermekimab) OR Placebo; Drug: MABp1 (Bermekimab)
- Placebo (Experimental)
  Interventions: Drug: MABp1 (Bermekimab) OR Placebo; Drug: MABp1 (Bermekimab)

INTERVENTIONS:
Drug: MABp1 (Bermekimab) OR Placebo — Period A: patients randomized 1:1 to weekly subcutaneous treatment with 400mg Bermekimab or matched Placebo for 12 weeks
Drug: MABp1 (Bermekimab) — Period B: all patients treated weekly with subcutaneous 400mg Bermekimab for 12 weeks

SUMMARY:
This is a proof-of concept RCT trying to generate evidence that inhibition of IL-1α through the administration of bermekimab may inhibit progression of SSc.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc also known as scleroderma) is a devastating chronic immune-mediated inflammatory syndrome that is characterized by progressive organ dysfunction. The most common affected systems are the skin, the gastrointestinal tract, the lungs and the heart. Capillary endothelium is involved leading to ischemia and digital necrosis. Patients develop an interstitial lung disease (ILD) prototype dominated by pulmonary hypertension (PHA) and failed gad exchange. Almost all patients are also presenting with signs of intestinal dysmotility leading to gastrointestinal reflux and bloating1. Hallmarks of SSc are fibrosis of the skin and internal organs, production of autoantibodies and vasculopathy. SSc is the only rheumatic disorder accompanied by substantial lethality; so far no specific treatment targeting the mechanism of pathogenesis is available.

The major denominator in the pathogenesis of SSc is the activation of fibroblast proliferation for the production of pre-collagen and the deposition of collagen in tissues; this leads to organ fibrosis and organ dysfunction. Activation of fibroblasts may come from transforming growth factor-β (TGFβ) and from interleukin (IL)-1α3. Circulating IL- 1α was measured in 66 Japanese patients with SSc and compared to 19 well-matched for age and gender healthy comparators. IL-1α was significantly greater than comparators; levels were similar between patients with limited cutaneous SSc and diffuse cutaneous SSc4. Contrary to IL-1β, IL-1α localizes on cell membranes and it is transported to the nucleus where it acts as a transcription factor. Whereas fibroblasts of healthy subjects produce IL-1α only after activation, fibroblasts from patients with SSc produce IL-1α extensively through a vicious autocrine pathway. More precisely, the IL-1R1 receptor is over-activated on fibroblasts from patients with SSc; this receptor binds to constitutively over-produced IL-1α by the same fibroblasts and this leads to a vicious cycle of fibroblast activation and production of pre-collagen4. Moreover, excess release of preformed IL-1α from the cytosol of damaged or stressed- cells leads to the recruitment of hematopoietic cells to the site of the inflammation through endothelial activation and disruption of the vascular wall5 explaining, at least in part, the vasculopathy of SSc. It has recently been shown that platelet microparticles and danger-associated molecular patterns (DAMPs) like high mobility group box-1 (HMGB1) are increased in the circulation of patients with SSc5. DAMPs can also prime platelet activation through an IL-1 dependent mechanism in patients with SSc The above evidence suggests that targeting IL-1α may be a novel target for the management of SSc.

Bermekimab (MABp1) is a first-in-class true human monoclonal antibody cloned directly from human B lymphocytes that specifically targets and neutralizes IL-1α. The drug has been tested so far in three randomized clinical trials (RCTs) in disease areas; metastatic colon carcinoma and hidradenitis suppurativa (HS). HS is a chronic devastating skin disorder that affects skin areas rich in apocrine glands. Bermekimab was administered intravenously every other week at a dose of 7.5mg/kg for 12 weeks; efficacy was compared to placebo. A total of 20 patients with severe HS who have failed or who were not eligible for adalimumab treatment were enrolled in this RCT; 60% responded to bermekimab compared to 10% of placebo comparators (p: 0.035). The salient feature of this trial was the provision of a proof-of-concept for the mechanism of action of bermekimab involving the down-regulation of the production of human β-defensin-2 (hBD-2). More precisely, whole blood was stimulated at the end of the 12-week treatment period with heat-killed Staphylococcus aureus. The total blood capacity of placebo-treated comparators was negatively associated with the decrease of the involved skin depth as measured by ultrasound; this negative association ceased to exist among bermekimab-treated patients. In another large- scale RCT , bermekimab was intravenously administered in 207 patients with metastatic or unresectable colorectal cancer and compared with 102 patients treated with placebo. The study primary endpoint was composite involving stable or increased lean body mass and stability or improvement in at least two or three symptoms of pain, fatigue and anorexia. This was achieved in 33% of bermekimab-treated and 19% of placebo-treated patients respectively (p: 0.0045).

ELIGIBILITY:
INCLUSION CRITERIA

* Age more than or equal to 18 years
* Both genders
* In the case of women of childbearing age, an adequate method of contraception should be used during the study. Contraception should be maintained at least until discontinuation of treatment. Prior to admission to the study, a pregnancy test will be performed to exclude pregnancy.
* Written informed consent
* Definite classification into SSc according to American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) criteria
* Modified Rodnan Skin Score (mRSS) units more than or equal to 15 and less than 40

EXCLUSION CRITERIA

* Age less than 18 years
* Denial to consent
* Pregnancy or lactation
* Renal crisis by SSc
* Major surgery the last 4 weeks prior to screening
* Known hypersensitivity to human, humanized, or murine monoclonal antibodies
* Active tuberculosis defined by the intake of drugs for recent tuberculosis
* Latent tuberculosis as defined by the positive interferon-γ releasing assay (IGRA)
* Chronic infection by the human immunodeficiency virus (HIV)
* Any primary immunodeficiency
* Hepatic dysfunction defined as aspartate aminotransferase more than 5 times the upper normal limit (UNL) or total bilirubin more than 5 times the UNL
* Any active bacterial infection
* Active solid tumor or hematologic malignancy
* Malabsorption requiring total parenteral nutrition
* Neutropenia defined as any absolute neutrophil count lower than 1,000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Score of inhibition of SSc progression | 2 years
  A positive score will comprise at least four of the following evaluation elements.
  * At least 30% decrease of the number of inflamed joints
  * At least 30% decrease of the number of digital ulcers
  * At least 30% decrease of the mRSS
  * At least 50% decrease of the UCLA GIT scoring system
  * At least 50% increase of the SF-36
  * At least 50% decrease of VAS for SSc
  * At least 50% decrease of VAS for fatigue
  * At least 50% decrease of VAS for dyspnea
  * Any increase of BMI ( kg/m2 )
  * Any increase of carbon monoxide diffusing capacity (DLCO)
  * Any increase of forced vital capacity (FVC)
  * At least 10% increase of the left ventricle ejection fraction (LVEF)
  * At least 10% decrease of the pulmonary artery pressure
  * At least 10% decrease of the capillary density as assessed by NCMT

SECONDARY OUTCOMES:
Secondary endpoints | 2 years
  The change of the achievement of a positive score of inhibition of SSc progression at week 24 compared to week 12 among patients originally allocated from week 0 to the bermekimab arm The change of the achievement of a positive score of inhibition of SSc progression at week 24 compared to week 12 among patients originally allocated from week 0 to the placebo arm The comparison of the score of inhibition of SSc progression at week 24 between the two groups of treatment The change of each of the elements of the score of inhibition of SSc progression at week 12 between the two groups of treatment. Comparisons for all qualitative variables of the secondary endpoints will be done by the Fisher exact test. Odds ratio and 95% confidence intervals will be calculated according to Mantel and Haenszel's statistics. Comparisons for all quantitative variables of the secondary endpoints will be done by non-parametric statistics.

OTHER OUTCOMES:
Endothelin-1 | 2 years
  Comparative kinetics of endothelin-1 between the two groups of treatment.
VEGF | 2 years
  Comparative kinetics of VEGF between the two groups of treatment.
TGFβ | 2 years
  Comparative kinetics of TGFβ between the two groups of treatment.
Pro-BNP | 2 years
  Comparative kinetics of pro-BNP between the two groups of treatment.
HMGB1 | 2 years
  Comparative kinetics of HMGB1 between the two groups of treatment.
IL-1α | 2 years
  Comparative kinetics ofIL-1α between the two groups of treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Department of Pathophysiology, LAIKO Athens General Hospital, Athens, Attica
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens, Attica

IPD SHARING:
Plan to Share IPD: No